CLINICAL TRIAL: NCT00720291
Title: Inflammation and Treatment of Bacterial Vaginosis Near Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Heather Norton, MD, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR # 17069
Record Dates: First submitted 2008-02-19; First posted 2008-07-22 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2010-01

CONDITIONS: Bacterial Vaginosis
Keywords: Metronidazole; BV; Pregnancy
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole (Active Comparator): Subjects who are randomly assigned to receive metronidazole 500 mg po for a period of 7 days following diagnosis of asymptomatic BV.
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Subjects who are randomly assigned to receive a placebo for a period of 7 days following the diagnosis of asymptomatic BV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — Patients who are randomly assigned to receive Metronidazole will receive 500 mg po bid Metronidazole for 7 days
  Other Names: Flagyl, CAS# 443-48-1
  Arms: Metronidazole
Drug: Placebo — Patients who are randomly assigned to receive a placebo will receive a placebo pill po bid for 7 days.
  Arms: Placebo

SUMMARY:
Most studies demonstrate that untreated bacterial vaginosis increases the rate of preterm birth. Despite this, there is no evidence that screening and treatment of asymptomatic bacterial vaginosis nor interpregnancy treatment of endometritis decreases the subsequent rate of preterm birth. However, treatment of symptomatic bacterial vaginosis has been associated with a modest reduction in subsequent preterm birth. Potential mechanisms for this reduction include a decrease in peripheral maternal pro-inflammatory activation of the TH1 inflammatory cascade with treatment, however this direct pathway has not been elucidated. The approved treatment for bacterial vaginosis during pregnancy consists of Metronidazole 500mg BID for 7 days. A more complete understanding of the effect of Metronidazole on maternal inflammation would be useful in designing strategies to reduce the rates of preterm birth.

This study proposes to determine the effect of standard treatment of BV carriage on maternal serum markers of inflammation. This will be accomplished by giving patients with asymptomatic BV either the standard treatment of metronidazole or a placebo for 7 days. Blood will be drawn to compare levels of Interleukins 1 and 6 as well as Tumor Necrosis Factor Alpha.

ELIGIBILITY:
Inclusion Criteria:

* 32 weeks gestation or greater
* Multiparity
* No history of preterm birth
* English speaking
* Ability to provide informed consent
* Bacterial vaginosis by gram stain

Exclusion Criteria:

* Acute infections at any site
* Active autoimmune disease
* Current anti-inflammatory use
* Symptomatic bacterial vaginosis
* Previous adverse reaction to metronidazole
* Reports ongoing ethanol consumption

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2010-11-23 (Actual); Study Completion 2010-11-23 (Actual)

PRIMARY OUTCOMES:
Levels of Interleukins 1 and 6 as well as Tumor Necrosis Factor Alpha | 3-5 days after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Heather Norton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States